CLINICAL TRIAL: NCT01644019
Title: Prehospital Telemedical Support in Acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005-1003-0034-2; PtJ-Az.: z0909im002b (Other Grant/Funding Number: PTJ)
Record Dates: First submitted 2012-07-12; First posted 2012-07-18 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Acute Stroke
Keywords: stroke; teleconsultation; telemedicine; emergency medical service
MeSH Terms: conditions — Stroke | interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device: Teleconsultation (Experimental): In cases of suspected acute stroke (including intracranial hemorrhage), if patients give informed consent the paramedics can use this system to contact a so called "tele-EMS physician" who has an audio-connection to the EMS team and receives vital parameters (e.g., ECG, pulse oximetry, non-invasive blood pressure) in real-time. The transmission of still pictures (taken with a smartphone), 12-lead-ECGs and video streaming from the inside of the ambulance can also be carried out, if indicated. The tele-EMS physician supports the EMS team in obtaining all relevant medical history, neurological diagnosis, general diagnosis and can delegate the application of medications. This can be carried out to bridge the time to the arrival of an EMS physician or in less severe cases without an EMS physician on-scene. The quality of prehospital care and the possible influences on the initial inhospital phase should be investigated and compared with regular EMS.
  Interventions: Procedure: Teleconsultation

INTERVENTIONS:
Procedure: Teleconsultation — Teleconsultation of an EMS physician in cases of suspected acute stroke

SUMMARY:
The aim of the study is to investigate the quality of prehospital emergency care in acute stroke, when paramedics are supported telemedically by an EMS physician.

DETAILED DESCRIPTION:
Six ambulances from five different Emergency Medical Service (EMS) districts are equipped with a portable telemedicine system. In cases of suspected acute stroke (including intracranial hemorrhage), the paramedics can use this system to contact a so called "tele-EMS physician" after consent of the patient is obtained. The tele-EMS physician has an audio-connection to the EMS team and receives vital parameters (e.g., ECG, pulse oximetry, non-invasive blood pressure) in real-time. The transmission of still pictures (taken with a smartphone), 12-lead-ECGs and video streaming from the inside of the ambulance can also be carried out, if indicated. The tele-EMS physician supports the EMS team in obtaining all relevant medical history, neurological diagnosis, general diagnosis and can delegate the application of medications. This can be carried out to bridge the time to the arrival of an EMS physician or in less severe cases without an EMS physician on-scene. The quality of prehospital care and the possible influences on the initial inhospital phase should be investigated and compared with regular EMS.

ELIGIBILITY:
Inclusion Criteria:

* suspected acute stroke
* verbal consent for teleconsultation obtained or patient is not able to consent due to the severity of the emergency

Exclusion Criteria:

* no suspected stroke
* patient refuses consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Quality of prehospital care | average 1 hour
  Analysis of the quality of prehospital care on the basis of published guidelines for acute stroke

SECONDARY OUTCOMES:
Clinical time intervals | 12 hours
  Prehospital and in-hospital time intervals: on-scene-time, contact to hospital time, door (hospital) to cerebral imaging, door (hospital) to thrombolysis
Diagnostic quality | up to 28 days
  Comparison of prehospital and definitive diagnosis
Information transfer | 2 hours
  Amount of stroke specific information that is transferred to the admitting hospital.
choice of appropriate hospital | average 1 hour
  Evaluation how many patients are transported to an appropriate facility (stroke unit)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Rossaint, Prof. Dr., Study Chair — University Hospital Aachen, Germany, Department of Anesthesiology; Jörg C Brokmann, Dr., Principal Investigator — University Hospital Aachen, Germany, Emergency Department
Locations (1):
- University Hospital Aachen, Aachen, Germany